CLINICAL TRIAL: NCT03404115
Title: A Multi-Center, Phase 2b, Randomized, Double Masked, Parallel-Group, Vehicle-Controlled, Clinical Study to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solution (0.25% and 0.1%) Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: A Multi-Center, Randomized, Double Masked, Parallel-Group, Vehicle-Controlled, Clinical Study to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solution in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-DED-009
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2023-01

CONDITIONS: Dry Eye Syndrome
Keywords: reproxalap
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Reproxalap Ophthalmic Solution (0.25%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Reproxalap Ophthalmic Solution (0.1%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.1%)
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered for approximately twelve weeks.
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Reproxalap Ophthalmic Solution (0.1%) — Reproxalap Ophthalmic Solution (0.1%) administered for approximately twelve weeks.
  Arms: Reproxalap Ophthalmic Solution (0.1%)
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution administered for approximately twelve weeks.
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
A Multi-Center, Phase 2b, Randomized, Double Masked, Parallel-Group, Vehicle-Controlled, Clinical Study to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solution (0.25% and 0.1%) Compared to Vehicle in Subjects with Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age of either gender and any race;
* Have a reported history of dry eye for at least 6 months prior to Visit 1;
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1;

Exclusion Criteria:

* Have any clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have used any eye drops within 2 hours of Visit 1;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Have used cyclosporine 0.05% or lifitigrast 5.0% ophthalmic solution within 90 days of Visit 1;
* Have any planned ocular and/or lid surgeries over the study period or any ocular surgery within 6 months of Visit 1;
* Be using or anticipate using temporary punctal plugs during the study that have not been stable within 30 days of Visit 1;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - The Eye Care Group, Waterbury, Connecticut
  - Midwest Cornea Associates, Indianapolis, Indiana
  - Central Maine Eye Care, Lewiston, Maine
  - Andover Eye Associates, Andover, Massachusetts
  - Andover Eye Associates, Raynham, Massachusetts
  - Total Eye Care, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clark D, Sheppard J, Brady TC. A Randomized Double-Masked Phase 2a Trial to Evaluate Activity and Safety of Topical Ocular Reproxalap, a Novel RASP Inhibitor, in Dry Eye Disease. J Ocul Pharmacol Ther. 2021 May;37(4):193-199. doi: 10.1089/jop.2020.0087. Epub 2021 Jan 15. PMID 33450164

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.1%) | Vehicle Ophthalmic Solution
Started | 100 | 100 | 100
Completed | 97 | 88 | 99
Not Completed | 3 | 12 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.1%) | Vehicle Ophthalmic Solution | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 58 | 50 | 51 | 159
  >=65 years | 42 | 50 | 49 | 141
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 28 | 179
  Male | 25 | 24 | 72 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 1 | 7
  Not Hispanic or Latino | 98 | 96 | 99 | 293
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 22 | 17 | 17 | 56
  White | 77 | 80 | 80 | 237
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 100 | 300
Iris Color (Right Eye) [Count of Participants; unit: Participants]
  Black | 1 | 1 | 2 | 4
  Blue | 15 | 22 | 26 | 63
  Brown | 55 | 47 | 46 | 148
  Green | 7 | 11 | 10 | 28
  Hazel | 22 | 17 | 16 | 55
  Gray | 0 | 2 | 0 | 2
  Other | 0 | 0 | 0 | 0
Iris Color (Left Eye) [Count of Participants; unit: Participants]
  Black | 1 | 1 | 2 | 4
  Blue | 15 | 22 | 26 | 63
  Brown | 55 | 47 | 46 | 148
  Green | 7 | 11 | 10 | 28
  Hazel | 22 | 17 | 16 | 55
  Gray | 0 | 2 | 0 | 2
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of ADX-102 on the Ora Calibra® Discomfort & 4-Symptom Questionnaire for Dryness.
Description: Change from baseline comparison of ADX-102 to Vehicle on the Ora Calibra® Discomfort & 4-Symptom Questionnaire (0 = least, 5 = most) for dryness across all time points. The intervention was administered bilaterally. The Least Squares Mean (Standard Error) was derived from Mixed Model Repeated Measure for change from baseline calculated using baseline score, visit, treatment, and visit-by-treatment interaction.
Time Frame: Efficacy assessment period (Day 1 through Day 85) - assessed on Days 1, 15, 29, 57, and 85.
Population: Intent to treat population with observed data only.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Reproxalap (0.25%): Reproxalap Ophthalmic Solution (0.25%): Reproxalap Ophthalmic Solution (0.25%) administered for approximately twelve weeks.
- Reproxalap (0.1%): Reproxalap Ophthalmic Solution (0.1%): Reproxalap Ophthalmic Solution (0.1%) administered for approximately twelve weeks.
- Vehicle: Vehicle Ophthalmic Solution: Vehicle Ophthalmic Solution administered for approximately twelve weeks.
Arm/Group | Reproxalap (0.25%) | Reproxalap (0.1%) | Vehicle
Number analyzed (Participants) | 100 | 100 | 100
units on a scale | -0.7 (0.09) | -0.5 (0.08) | -0.4 (0.08)

ADVERSE EVENTS:
Time Frame: The period of time when adverse events were collected was approximately 3 months.
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) | Reproxalap Ophthalmic Solution (0.1%) | Vehicle Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 1/100 | 1/100 | 0/100
Other Adverse Events (participants affected / at risk) | 93/100 | 37/100 | 2/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap Ophthalmic Solution (0.25%) (N=100) | Reproxalap Ophthalmic Solution (0.1%) (N=100) | Vehicle Ophthalmic Solution (N=100)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 — The serious adverse event of angina pectoris was deemed not related to study drug.
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 — The serious adverse event of vertigo was deemed unlikely to be related to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap Ophthalmic Solution (0.25%) (N=100) | Reproxalap Ophthalmic Solution (0.1%) (N=100) | Vehicle Ophthalmic Solution (N=100)
General disorders and administration site conditions (General disorders) | 93 | 37 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT03404115/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT03404115/SAP_001.pdf